CLINICAL TRIAL: NCT05320276
Title: Redictors of Non-accESs to therapeutiC EducAtion Programs Among Patients With Type 2 Diabetes, and/or Asthma, and/or Chronic Heart Failure in an Emergency Setting
Brief Title: Predictors of Non-accESs to therapeutiC EducAtion Programs Among Patients With Type 2 Diabetes, and/or Asthma, and/or Chronic Heart Failure in an Emergency Setting
Acronym: ESCAPE
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: ESCAPE
Record Dates: First submitted 2022-03-31; First posted 2022-04-11 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Therapeutic Education Program; Emergencies; Diabetes; Asthma; Heart Failure
MeSH Terms: conditions — Emergencies; Diabetes Mellitus; Asthma; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chronic diseases are frequent and potentially severe. Type II diabetes, asthma and heart failure affect 3.3 million, 4 million and 1 million people respectively in France. They are sources of avoidable mortality as well as disabilities leading to a loss of years of full health life (DALYS). Cumulatively, they were responsible for the loss of more than 1 million DALYS in 2019 in France. National and international recommendations also include TVE in the management of these three diseases.

This severity can be reduced by better management underpinned by therapeutic education. By improving their knowledge of the disease, it allows a better adherence of patients to the care project, the achievement of clinical and biological objectives, a decrease in the number of emergency room visits and unscheduled hospitalizations, and an improvement in the quality of life during the course of three frequent chronic diseases such as type 2 diabetes, asthma and heart failure.

However, participation in a therapeutic education program remains highly variable depending on many parameters. Lack of information seems to play a major role in this context.

In the Ile de France region, the density of available TEP programs is high, particularly in Paris. The three chronic diseases that are managed by an advanced practice nurse with a PCS mention have the largest number of TVE programs in Paris: type 2 diabetes (32, and 6 for diabetic foot), asthma and heart failure.

In an urban area with a good supply of TVE facilities, how can investigators explain the lack of integration of these facilities into the care pathway? Among the diverse patient population consulting an emergency department suffering from type II diabetes, asthma or heart failure, investigators wish to determine the proportion of patients who have not been offered TVE during their care.

Investigators will then try to identify demographic, socioeconomic, and medical factors statistically associated with the absence of FTE proposal.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age is ≥ 18 years
* Patient consulting the GHPSJ emergency department for any reason
* Patient with a chronic disease among type 2 diabetes and/or asthma and/or heart failure
* Francophone patient

Exclusion Criteria:

* Diagnosis of the chronic disease in the context of its current management in the emergency room
* Patient being followed outside of Ile de France for the chronic disease studied
* Patient with dementia or cognitive disorders
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under legal protection
* Patient opposing the use of his data for this research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients visit the emergency department for any reason between 12/15/2021 and 3/30/2022 and have at least one of the following chronic conditions: type 2 diabetes, asthma or heart failure.
Sampling Method: Non-Probability Sample
Enrollment: 297 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
Frequency of patients with chronic diseases seen in the emergency department who have not been offered an educational program | Day 1
  This outcome corresponds to the number of patients who have not been offered participation in a therapeutic education program during their course of care since the diagnosis of their chronic disease.

SECONDARY OUTCOMES:
Patient Characteristics Associated with Not Offering a Therapeutic Education Program During the Course of Care | Day 1
  This outcome corresponds to the demographic, social, economic and medical characteristics statistically associated with the absence of a therapeutic education proposal.
Identification of reasons for refusal to participate | Day 1
  This outcome corresponds to the reason for declining to participate in an TEP program for patients who have been offered one.

CONTACTS AND LOCATIONS:
Overall Officials: Camille GERLIER, MD, Principal Investigator — Groupe Hopsitalier Paris Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Background] Odgers-Jewell K, Ball LE, Kelly JT, Isenring EA, Reidlinger DP, Thomas R. Effectiveness of group-based self-management education for individuals with Type 2 diabetes: a systematic review with meta-analyses and meta-regression. Diabet Med. 2017 Aug;34(8):1027-1039. doi: 10.1111/dme.13340. Epub 2017 Mar 20. PMID 28226200
- [Background] McGhan SL, Cicutto LC, Befus AD. Advances in development and evaluation of asthma education programs. Curr Opin Pulm Med. 2005 Jan;11(1):61-8. doi: 10.1097/01.mcp.0000146783.18716.31. PMID 15591890
- [Background] Rice H, Say R, Betihavas V. The effect of nurse-led education on hospitalisation, readmission, quality of life and cost in adults with heart failure. A systematic review. Patient Educ Couns. 2018 Mar;101(3):363-374. doi: 10.1016/j.pec.2017.10.002. Epub 2017 Oct 5. PMID 29102442
- See also: Related Info — https://www.em-consulte.com/article/1196953/competences-attendues-de-l-infirmiere-de-pratique-